CLINICAL TRIAL: NCT00908297
Title: Safety, Tolerability and Efficacy of Coenzyme Q10 in Hemodialysis Patients: Aim 1
Brief Title: Safety and Tolerability of Coenzyme Q10 in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jonathan Himmelfarb, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 35580-D; R21AT004265-01A2 (NIH)
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Disease; End Stage Renal Disease; Atherosclerosis; Oxidative Stress
Keywords: Cardiovascular disease; End stage renal disease; Atherosclerosis; Oxidative stress; Antioxidants
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Failure, Chronic; Atherosclerosis | interventions — coenzyme Q10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — By mouth (wafer) once daily for duration of study (8 weeks).
  Dose escalation:
  * 300 mg for two weeks
  * 600 mg for two weeks
  * 1200 mg for two weeks
  * 1800 mg for final two weeks
  Other Names: CoQ10

SUMMARY:
The purpose of this study is to determine the safety and tolerability of the dietary supplement Coenzyme Q10 in hemodialysis patients.

DETAILED DESCRIPTION:
There are more than 400,000 patients receiving dialysis in the United States, and we expect that this number will go up. For those on hemodialysis, cardiovascular disease (CVD) accounts for a large part of the health problems that these patients have. Cardiovascular problems come from damage to the heart or blood vessels.

At present, we have no treatments proven to help prevent CVD in those on dialysis. For the general population, we know about many factors that increase the risk of CVD, such as having a high level of "bad" cholesterol. But for people on dialysis, we believe that there are other risk factors that are just as important in the development of CVD.

People on dialysis often have high blood levels of waste products. This is called "uremia". We believe that uremia can set up chemical reactions in the blood which can lead to hardening of the arteries (atherosclerosis), an important part of CVD. Compounds called antioxidants, which stop the chemical reactions, may help prevent CVD.

Coenzyme Q10 is a naturally occurring compound in blood and tissues. It is also a readily available dietary supplement often used as an alternative and complementary medicine. It is a powerful antioxidant. Previous studies have shown that blood levels of coenzyme Q10 are decreased in hemodialysis patients. Because of this, it is important for us to find out if giving coenzyme Q10 to hemodialysis patients can help prevent CVD. However, at present, there are no studies which carefully look at the safety and tolerability of coenzyme Q10, and whether it helps stops the harmful chemical reactions in the blood.

In addition, many people take medications called "statins" to help reduce risk for cardiovascular disease. We know that statins can lower coenzyme Q10. It is important for us to know if hemodialysis patients taking statins have lower levels of coenzyme Q10. It may be that therapy with coenzyme Q10 could increase the beneficial effects of statin therapy in hemodialysis patients.

In this study, we will test to see if different doses of the dietary supplement coenzyme Q10 will be safe and well tolerated in hemodialysis patients. This is with a view to later studies to determine if coenzyme Q10 will help stop harmful chemical reactions in the blood for hemodialysis patients. This study will help us prepare for future studies of coenzyme Q10, by demonstrating the safely and tolerability of this compound in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage renal disease receiving thrice weekly hemodialysis
* Age > 18 and < 85 years
* Life expectancy greater than one year
* Ability to understand and provide informed consent for participation in the study
* Mean baseline plasma F2-isoprostane concentration > 50 pg/mL

Exclusion Criteria:

* History of poor adherence to hemodialysis or medical regimen
* Prisoners, patients with significant mental illness, and other vulnerable populations
* AIDS (HIV seropositivity is not an exclusion criteria)
* Active malignancy excluding basal cell carcinoma of the skin
* Gastrointestinal dysfunction requiring parenteral nutrition
* History of functional kidney transplant < 6 months prior to study entry
* Anticipated live donor kidney transplant
* Patients taking vitamin E supplements > 60 IU/day, vitamin C > 50 mg/day or other antioxidant or nutritional supplements
* Incident hemodialysis patients (defined as within 90 days of dialysis initiation)
* Patients hospitalized within the past 60 days
* Patients being dialyzed with a tunneled catheter as a temporary vascular access
* Patients with a history of a major atherosclerotic event (defined as combined incidence of myocardial infarction, urgent target-vessel revascularization, coronary bypass surgery, and stroke) within six months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety Measures: * Laboratory tests on serum: Comprehensive metabolic panel and creatinine phosphokinase. * Electrocardiogram, physical examination findings, and adverse events. | Every two weeks
Efficacy Measures: Markers in the blood indicating "oxidative stress" | Every two weeks

SECONDARY OUTCOMES:
Serum biomarkers of Cardiovascular condition and health | At baseline study visit and last study visit

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Himmelfarb, MD, Principal Investigator — University of Washington - Kidney Research Institute
Locations (1):
- Northwest Kidney Centers - Scribner, Seattle, Washington, United States

REFERENCES:
- [Derived] Yeung CK, Billings FT 4th, Claessens AJ, Roshanravan B, Linke L, Sundell MB, Ahmad S, Shao B, Shen DD, Ikizler TA, Himmelfarb J. Coenzyme Q10 dose-escalation study in hemodialysis patients: safety, tolerability, and effect on oxidative stress. BMC Nephrol. 2015 Nov 3;16:183. doi: 10.1186/s12882-015-0178-2. PMID 26531095
- See also: Northwest Kidney Centers — http://www.nwkidney.org/